CLINICAL TRIAL: NCT06190626
Title: Longitudinal Prospective Natural History Study of Retinopathy in Zellweger Spectrum Disorder
Acronym: ZSDvision
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Nancy Braverman, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2024-9679
Record Dates: First submitted 2023-12-04; First posted 2024-01-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Zellweger Spectrum Disorder
Keywords: ZSD; PEX gene mutation; Retinopathy
MeSH Terms: conditions — Zellweger Syndrome; Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to define the course of the retinal degeneration in a ZSD patient cohort.

The objective of this study is to gather information so the investigators can:

1. define the course of the retinal degeneration in a ZSD patient cohort with retinal degeneration
2. define what tests best monitor the progression of the retinal degeneration
3. generate prognostic information about vision loss in ZSD.

At each yearly visit, the participants will answer a functional vision questionnaire, have a physical evaluation, blood test, and participate in a variety of vision tests. The investigators will also collect pertinent medical history.

Participants will travel to study site. The study will provide financial support for board and travel.

DETAILED DESCRIPTION:
Participants/guardians will have a 1-hour virtual interview before the first visit to review the tests and determine which tests the participant is able to perform.

Below is a list of the vision tests used for this study:

Prior to each visit, the participant will complete the PedEyeQ or VFQ-25 questionnaire about functional vision.

At each clinic visit :

* Refraction and glasses test: this is a general vision test, as commonly conducted by an optometrist, before and after pupil dilation
* Best corrected visual acuity: the participant's vision will be tested using cards or a chart.
* Contrast sensitivity: the participant's ability to detect contrast will be tested using a chart.
* Visual field: the participant's field of vision will be tested by asking them to indicate when they see a stimulus.
* Reading test: the participant's ability to see written text will be tested using the International Reading Speed Test
* Color vision test: the participant's ability to see color will be tested using cards
* Eye exam: the participant's eyes will be examined with a lamp
* Pupil dilation: to allow the completion of some tests, the participant's pupils will be dilated using medicated eye drops
* Microperimetry: the participant's macula (central retina) will be visualized.
* Fundus photography: the participant's fundus (central retina) will be photographed in light and dark conditions
* Full field stimulus threshold test: the participant's ability to perceive light in different parts of their visual field will be tested
* Optical coherence tomography (OCT): detailed images of the participant's retina will be taken
* Fundus autofluorescence: the participant's retinal health will be assessed by imaging the natural fluorescent properties of their retinal pigment epithelium
* Chromatic pupillometry: the function of different cells in the participant's retina will be determined by measuring their response to light
* Multi-luminance mobility test (MLMT): the participant will walk through an obstacle course at varying light levels to test their functional vision in different light conditions.
* Blood collection: a blood sample will be collected and banked to measure peroxisome functions.

ELIGIBILITY:
Inclusion Criteria:

* confirmed ZSD with deleterious variants in PEX genes identified
* confirmed or expected retinal involvement

Exclusion Criteria:

* unable to perform a minimum of one vision test
* severe ZSD disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: any age, with appropriate diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with disease progression | 5 years
  Using various tests of vision measured annually, a description of disease progression will be defined in each participant.
Number of participants with common patterns of retinal degeneration observed | 5 years
  Vision test results from participants will be reviewed together to describe common patterns of retinal degeneration observed.

SECONDARY OUTCOMES:
Rate of progression of retinal degeneration | 5 years
  Statistical analysis using the data from Outcome 1, will be used to generate rate of progression per year over 5 years in each individual.
Correlation of rate retinal degeneration to age and overall ZSD disease severity | 5 years
  Statistical analysis using the data from Outcome 1, will be used to correlate rate of progression per year over 5 years to age and overall ZSD disease severity in each individual.
rate of progression of retinal degeneration | 5 years
  Statistical analysis using the data from Outcome 1, will be used to define variance between participants in rate of progression of retinal degeneration.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Braverman, MD, MS, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (3):
- University of Rochester Medical Center/Flaum Eye Institute, Rochester, New York, United States
- Canada (2):
  - Eye Institute of Alberta, Edmonton, Alberta
  - Research Institute-McGill University Health Center, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braverman NE, Raymond GV, Rizzo WB, Moser AB, Wilkinson ME, Stone EM, Steinberg SJ, Wangler MF, Rush ET, Hacia JG, Bose M. Peroxisome biogenesis disorders in the Zellweger spectrum: An overview of current diagnosis, clinical manifestations, and treatment guidelines. Mol Genet Metab. 2016 Mar;117(3):313-21. doi: 10.1016/j.ymgme.2015.12.009. Epub 2015 Dec 23. PMID 26750748
- [Background] Yergeau C, Coussa RG, Antaki F, Argyriou C, Koenekoop RK, Braverman NE. Zellweger Spectrum Disorder: Ophthalmic Findings from a New Natural History Study Cohort and Scoping Literature Review. Ophthalmology. 2023 Dec;130(12):1313-1326. doi: 10.1016/j.ophtha.2023.07.026. Epub 2023 Aug 2. PMID 37541626